CLINICAL TRIAL: NCT05330195
Title: The Effects of Bicycle Training on Gait and Balance in Children With Duchenne Muscular Dystrophy
Brief Title: Bicycle Ergometer Training in Duchenne Muscular Dystrophy
Acronym: BETDMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Numan Bulut, Research Assistant (Assistant of neuromuscular disorders unit), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022008
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Bicycle training; Gait; Balance
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Block Randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Home exercise program Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do these for 3 to 5 days a week. Also, aerobic training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 40 minutes total duration consisting of 5 min warm up and 5 min cool down period to children in treatment group
  Interventions: Other: Bicycle Ergometer Training; Other: Home-based exercise group
- Control Group (Active Comparator): Home Based Exercise Group Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do this program for 3-5 days a week.
  Interventions: Other: Home-based exercise group

INTERVENTIONS:
Other: Bicycle Ergometer Training — Bicycle ergometer training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 40 minutes total duration consisting of 5 min warm up and 5 min cool down period to children in treatment group.
  Arms: Treatment Group
Other: Home-based exercise group — Children will be given a home program including stretching, breathing, normal joint movement, body weight and mildly resistant exercises, and children will be asked to do these for 3 to 5 days a week.

SUMMARY:
The progressive muscle weakness and contractures of the patients adversely affect their gait and balance. It is known that the disorder of the patients' balance and gait affects their functional capacity. The aim of this study is to examine the effects of bicycle ergometer training on gait and balance in children with Duchenne Muscular Dystrophy. Twenty-four children with DMD included in the study will be divided into two groups as home program and home program+bicycle ergometer training with block randomization method. Home program including stretching, respiratory, range of motion, posture and mild resistance exercise with body weight will be asked to apply 3-5 days a week for 12 weeks, aerobic training will be performed 3 days a week for 12 weeks at 60% of their maximum hearth rate with 40 minutes total duration consisting of 5 min warm up and 5 min cool down period. Gait and balance were evaluated with GAITrite and Bertec Balance Check Screener, successively. Assessments will be applied at pre-training and after 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Children have diagnosis of DMD confirmed by genetic analysis,
* Children can walk with unsupported.

Exclusion criteria:

* Children have undergone any surgery or suffered injury of the lower limbs,
* Children have severe contractures of lower limbs,
* Children have low cooperation
* Children have comorbid disease,
* Children were applied regular aerobic training such as bicycle training and hydrotherapy in last 6 months.

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Because DMD is X linked recessive disorder, this disorder is seen in male.
Enrollment: 23 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Step Time and Cycle Time(Gait) | 5 minutes
  The gait of patients with DMD was assessed by GAITrite (CIR Systems Inc., Franklin, New Jersey, USA) electronic walkway system, objective assessment of spatio-temporal characteristics of gait, at a self-selected speed for 3 times. With this walkway system, ambulation time (s) was evaluated.
Step Length, Stride Length and base of support (Gait) | 5 minutes
  The gait of patients with DMD was assessed by GAITrite (CIR Systems Inc., Franklin, New Jersey, USA) electronic walkway system, objective assessment of spatio-temporal characteristics of gait, at a self-selected speed for 3 times. With this walkway system,step length (cm), stride length (cm) and base of support (cm) were evaluated.
Single support, double support, swing phase and stance phase (Gait) | 5 minutes
  The gait of patients with DMD was assessed by GAITrite (CIR Systems Inc., Franklin, New Jersey, USA) electronic walkway system, objective assessment of spatio-temporal characteristics of gait, at a self-selected speed for 3 times. With this walkway system, single support, double support, swing phase and stance phase were stated as %.
Velocity (Gait) | 5 minutes
  The gait of patients with DMD was assessed by GAITrite (CIR Systems Inc., Franklin, New Jersey, USA) electronic walkway system, objective assessment of spatio-temporal characteristics of gait, at a self-selected speed for 3 times. With this walkway system, Velocity (cm/s) was evaluated.
Cadence (Gait) | 5 minutes
  The gait of patients with DMD was assessed by GAITrite (CIR Systems Inc., Franklin, New Jersey, USA) electronic walkway system, objective assessment of spatio-temporal characteristics of gait, at a self-selected speed for 3 times. With this walkway system, cadence (steps/min) was recorded.
Balance (rigid surface) | 10 minutes
  The balance plate system used to assess balance and degree of postural sway was the Bertec Balance Check Screener™ (BP5050 Bertec Co., Columbus, OH, USA). The system consists of a 20 × 20-inch platform at ground level connected to a computer. Postural sway, which measures the displacement of the center of gravity, was assessed on rigid surface, in 2 conditions (eyes opened-closed) and 2 directions (anteroposterior and mediolateral).
Balance (perturbated surface) | 10 minutes
  The balance plate system used to assess balance and degree of postural sway was the Bertec Balance Check Screener™ (BP5050 Bertec Co., Columbus, OH, USA). The system consists of a 20 × 20-inch platform at ground level connected to a computer. Postural sway, which measures the displacement of the center of gravity, was assessed on perturbated surface, in 2 conditions (eyes opened-closed) and 2 directions (anteroposterior and mediolateral).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No